CLINICAL TRIAL: NCT04664296
Title: Epidemiology of CoV-2 SARS Infections: Dynamics of Community Contamination in Children and Adults
Brief Title: COVID-19 - SARS-CoV-2 Community Contamination in Children and Adults (Dyn3CEA_Nosocor)
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1100
Record Dates: First submitted 2020-12-10; First posted 2020-12-11 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Infection Viral
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children: Hospitalized children, 0 to 17 years of age, 25 subjects, consecutive sample survey
  Interventions: Other: Review of medical patient file
- Adults: Hospitalized adults, 18 years and above, 50 matched subjects
  Interventions: Other: Phone call interview

INTERVENTIONS:
Other: Review of medical patient file — Review of medical patient file, including patient tracing, brief summary of the disease course, barrier gestures, social distancing.
  Groups: Children
Other: Phone call interview — less than 15 minutes phone call
  Groups: Adults

SUMMARY:
Unlike other respiratory viruses such as influenza and Respiratory Syncytial Virus (RSV) where the child is the essential reservoir and central vector of intrafamilial contamination, the child is likely to be a small player in the transmission of Severe Acute Respiratory Syndrome CoronaVirus 2 (SRAS-CoV2) infection. This study aims to describe the age category of the first contact, within 14 days before the appearance of the first symptoms of the index case in order to describe the age categories of this first contaminant, globally, in the group of children and finally in the group of adults. This work is intended to provide food for discussion and to justify the distancing and containment measures imposed on children when their isolation has a deleterious impact that has now been established for some children.

ELIGIBILITY:
Inclusion Criteria:

1. Children after hospitalized in Hospices Civils de Lyon with Polymerase Chain Reaction (PCR) positive SARS-CoV2,
2. Adults hospitalized in Hospices Civils de Lyon and included in the NOSO-COR study with matching criteria described below.

   * Matching will be performed on family age characteristics and on the period of contamination included in the containment period to minimize bias, and if possible frequency matching according to admission in Intensive Care Unit ICU/Pediatric Intensive Care Unit (PICU), and to family structure (n of children / n of adults in the family).

Exclusion Criteria:

1. Any patient suspected of nosocomial infection.
2. Any patient death during the Covid-19 infection.
3. Any adult patient without children living home.
4. Opposition to participate.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospital-based population of children and adults:
  * Hospitalized children, 0 to 17 years of age, 25 subjects, consecutive sample survey
  * Hospitalized adults, 18 years and above, 50 matched subjects
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2020-12-21 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Percentage of possible contaminants, adults, adolescents and children with Covid-19 | at inclusion
  To describe the age category of the 1st possible contaminant in the index case to show the preponderance of possible adult and adolescent contaminants in the SARS-Cov-2 contamination.
  Percentage of possible contaminants, adults, adolescents and children, in matched children and adults with Covid-19.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Reanimation Pediatrique, Lyon, Rhone, France